CLINICAL TRIAL: NCT00329901
Title: A Phase 3, Multi-Center, Observer Blind, Controlled, Randomized Study to Compare the Immunogenicity and Safety of the Concomitant Administration of a Combined Tetanus, Reduced Diphtheria, and Acellular Pertussis (Tdap) Vaccine and Chiron (Now Novartis) Meningococcal ACWY Conjugate Vaccine, With Either One Dose of Acellular Pertussis (Tdap) Vaccine, or One Dose of Chiron (Now Novartis) Meningococcal ACWY Conjugate Vaccine, in Healthy Subjects Aged 11-25 Years
Brief Title: Immunogenicity and Safety of the Concomitant Administration of a Tdap Vaccine and Meningococcal ACWY Conjugate Vaccine in Healthy Subjects Aged 11-25 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V59P11; 2005-005519-12 (EudraCT Number)
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningitis; healthy subject; vaccine
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tdap + MenACWY-CRM (Experimental): Subjects received Tdap and MenACWY-CRM vaccines concomitantly, in separate arms
  Interventions: Biological: Meningococcal ACWY conjugate vaccine (MenACWY-CRM); Biological: Combined tetanus, reduced diphtheria and acellular pertussis vaccine (Tdap)
- Tdap + saline (Experimental): Subjects received Tdap vaccine and saline (placebo) concomitantly, in separate arms
  Interventions: Biological: Combined tetanus, reduced diphtheria and acellular pertussis vaccine (Tdap); Biological: saline placebo
- MenACWY-CRM + saline (Experimental): Subjects received MenACWY-CRM vaccine and saline (placebo) concomitantly, in separate arms
  Interventions: Biological: Meningococcal ACWY conjugate vaccine (MenACWY-CRM); Biological: saline placebo

INTERVENTIONS:
Biological: Meningococcal ACWY conjugate vaccine (MenACWY-CRM)
  Arms: MenACWY-CRM + saline; Tdap + MenACWY-CRM
Biological: Combined tetanus, reduced diphtheria and acellular pertussis vaccine (Tdap)
  Arms: Tdap + MenACWY-CRM; Tdap + saline
Biological: saline placebo — 4.5 mg sodium chloride per 0.5 ml dose
  Arms: MenACWY-CRM + saline; Tdap + saline

SUMMARY:
Immunogenicity and Safety of the Concomitant Administration of a Tdap Vaccine and Meningococcal ACWY Conjugate Vaccine in Healthy Subjects Aged 11-25 Years

ELIGIBILITY:
Inclusion Criteria:

* Male and female 11-25 years old healthy subjects;
* who had received the primary immunization with a vaccine containing DT or Tdap antigens and a T, Td, or Tdap booster injection at least 5 years prior to study entry

Exclusion Criteria:

* previous ascertained or suspected disease caused by N. meningitidis
* previously been immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s)
* serious acute, chronic or progressive disease
* history of any anaphylaxis, serious vaccine reactions, or allergy to any vaccine component
* known or suspected impairment/alteration of immune function, either congenital or acquired

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1072 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Information Services, Study Chair — Novartis Vaccines & Diagnostics
Locations (14):
- Italy (14):
  - Andria
  - Catania
  - Chieti
  - Ferrara
  - Genova
  - Lanciano
  - Massafra
  - Modena
  - Novara
  - Palermo
  - Pieve Di Soligo (TV)
  - Roma
  - Sassari
  - Taranto

REFERENCES:
- [Result] Gasparini R, Conversano M, Bona G, Gabutti G, Anemona A, Dull PM, Ceddia F. Randomized trial on the safety, tolerability, and immunogenicity of MenACWY-CRM, an investigational quadrivalent meningococcal glycoconjugate vaccine, administered concomitantly with a combined tetanus, reduced diphtheria, and acellular pertussis vaccine in adolescents and young adults. Clin Vaccine Immunol. 2010 Apr;17(4):537-44. doi: 10.1128/CVI.00436-09. Epub 2010 Feb 17. PMID 20164251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 14 centers in Italy.
Pre-assignment Details: All enrolled subjects participated in the trial.
Groups:
- Tdap + MenACWY-CRM: Subjects received Tdap vaccine and MenACWY-CRM vaccine concomitantly, in separate arms
- Tdap + Saline: Subjects received Tdap vaccine and saline (placebo)concomitantly, in separate arms
Period: Overall Study
Arm/Group | Tdap + MenACWY-CRM | Tdap + Saline | MenACWY-CRM + Saline
Started | 361 | 354 | 357
Completed | 352 | 349 | 353
Not Completed | 9 | 5 | 4
Not completed — Withdrawal by Subject | 4 | 3 | 2
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Unable to classify | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics are summarized for all enrolled population
Groups:
- Total: Total of all reporting groups
Arm/Group | Tdap + MenACWY-CRM | Tdap + Saline | MenACWY-CRM + Saline | Total
Number analyzed (Participants) | 361 | 354 | 357 | 1072
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (3.4) | 14.1 (3.2) | 14.3 (3.2) | 14.3 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 164 | 165 | 518
  Male | 172 | 190 | 192 | 554

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With an Immune Response Against Diphtheria, Tetanus and Pertussis, When Tdap is Concomitantly Administered With MenACWY-CRM Compared to Tdap Given Concomitantly With Saline Placebo
Description: To demonstrate that the immunogenicity of one injection of Tdap vaccine, concomitantly administered with MenACWY-CRM vaccine, is not inferior to that of one injection of Tdap vaccine, concomitantly administered with saline placebo, in terms of
  1. the percentage of subjects with antibody levels against diphtheria toxin ≥ 1.0 IU/mL and against tetanus toxin ≥ 1.0 IU/mL and
  2. the percentage of subjects with at least 4 fold increase in antibody levels against pertussis toxin (PT), filamentous hemagglutinin (FHA) and pertactin (PRN) at 1 month after immunization, as measured by enzyme linked immunosorbent assay (ELISA).
Time Frame: 1 month after vaccination (Day 29)
Population: Analysis was done on the per-protocol population i.e all subjects who received all the relevant doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol violation as defined prior to unblinding
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- Tdap+MenACWY-CRM: Subjects received Tdap vaccine and MenACWY-CRM vaccine concomitantly, in separate arms
- Tdap+Saline: Subjects received Tdap vaccine and saline (placebo) concomitantly, in separate arms
Arm/Group | Tdap+MenACWY-CRM | Tdap+Saline
Number analyzed (Participants) | 350 | 345
Percentages of subjects
  Day 1 (diphtheria) | 4 [2 to 7] | 5 [3 to 7]
  Day 29 (diphtheria) | 94 [91 to 96] | 85 [80 to 88]
  Day 1 (tetanus ) | 25 [20 to 30] | 36 [31 to 42]
  Day 29 (tetanus ) | 100 [99 to 100] | 99 [98 to 100]
  Day 29 (PT) 4-fold increase (N=286, 287) | 76 [70 to 80] | 81 [76 to 85]
  Day 29 (FHA)4-fold increase (N=286, 287) | 83 [78 to 87] | 86 [82 to 90]
  Day 29 (PRN) 4-fold increase (N=285, 287) | 84 [79 to 88] | 91 [87 to 94]
Statistical Analysis 1: Comparison: Tdap+MenACWY-CRM vs Tdap+Saline; Non-inferiority of anti-diphtheria immune response following concomitant administration of Tdap with MenACWY-CRM as compared to Tdap given with placebo saline; Test type: Non-Inferiority or Equivalence — The immune response to Tdap + MenACWY-CRM was considered non-inferior to that of Tdap+saline if for all five antigens (diphtheria, tetanus, PT, FHA, PRN) the lower limit of the 95% CI of the difference [(Tdap + MenACWY-CRM) minus(Tdap + saline)] was greater than -10, at 1 month (Day 29) after vaccination; Vaccine Group difference = 9, 95% CI 2-sided [5 to 14]
Statistical Analysis 2: Comparison: Tdap+MenACWY-CRM vs Tdap+Saline; Non-inferiority of anti-tetanus immune response following concomitant administration of Tdap with MenACWY-CRM compared to Tdap given concomitantly with saline placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Vaccine Group Difference = 1, 95% CI 2-sided [-1 to 2]
Statistical Analysis 3: Comparison: Tdap+MenACWY-CRM vs Tdap+Saline; Non-inferiority of anti-PT antigen immune response following concomitant administration of Tdap with MenACWY as compared to Tdap given concomitantly with saline placebo; Test type: Non-Inferiority or Equivalence — The immune response to Tdap + MenACWY-CRM was considered non-inferior to that of Tdap+saline if for all five antigens (diphtheria, tetanus, PT, FHA, PRN) the lower limit of the 95% CI of the difference [(Tdap + MenACWY-CRM) minus (Tdap + saline)] was greater than -10, at 1 month (Day 29) after vaccination; Vaccine Group difference = -5, 95% CI 2-sided [-12 to 1]
Statistical Analysis 4: Comparison: Tdap+MenACWY-CRM vs Tdap+Saline; Non-inferiority of anti-FHA antigen immune response following concomitant administration of Tdap with MenACWY as compared to Tdap given concomitantly with saline placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; Vaccine Group Difference = -3, 95% CI 2-sided [-9 to 3]
Statistical Analysis 5: Comparison: Tdap+MenACWY-CRM vs Tdap+Saline; Non-inferiority of anti-PRN antigen immune response following concomitant administration of Tdap with MenACWY as compared to Tdap given concomitantly with saline placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; Vaccine Group Difference = -7, 95% CI 2-sided [-13 to -2]

2. Secondary Outcome: Percentage of Subjects With Anti-diphtheria and Anti-tetanus Concentrations ≥ 0.1 IU/mL When Tdap is Administered Concomitantly With MenACWY-CRM Vaccine Compared to Tdap Given Concomitantly With Saline Placebo
Description: The percentage of subjects with anti-diphtheria and anti-tetanus concentrations ≥ 0.1 IU/mL (as measured by ELISA) following concomitant administration of Tdap vaccine with MenACWY-CRM vaccine as compared to when Tdap was given concomitantly with saline placebo.
Time Frame: 1 month after vaccination (Day 29)
Population: Analysis was done on per-protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Tdap+MenACWY-CRM | Tdap+Saline
Number analyzed (Participants) | 350 | 345
Percentages of subjects
  Day 1 (diphtheria) | 55 [50 to 60] | 63 [57 to 68]
  Day 29 (diphtheria) | 100 [99 to 100] | 100 [98 to 100]
  Day 1 (tetanus) | 97 [95 to 99] | 97 [95 to 99]
  Day 29 (tetanus) | 100 [99 to 100] | 100 [99 to 100]

3. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies Against Diphtheria,Tetanus and Pertussis Antigens After Concomitant Administration of Tdap With MenACWY-CRM Compared to Tdap Given Concomitantly With Saline Placebo
Description: The geometric mean concentrations of antibodies ≥ 0.1 IU/mL against diphtheria, tetanus and pertussis (PT, FHA and PRN) antigens in subjects, as measured by ELISA, following concomitant administration of Tdap with MenACWY-CRM as compared to when Tdap given concomitantly with saline placebo.
Time Frame: 1 month after vaccination (Day 29)
Population: Analysis was done on per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- Tdap+ MenACWY-CRM: Subjects received Tdap vaccine and MenACWY-CRM vaccine concomitantly, in separate arms
Arm/Group | Tdap+ MenACWY-CRM | Tdap+Saline
Number analyzed (Participants) | 350 | 345
IU/mL
  Day 1 (diptheria) | 0.11 [0.085 to 0.14] | 0.12 [0.096 to 0.16]
  Day 29 (diptheria) | 7.96 [6.19 to 10] | 2.77 [2.15 to 3.57]
  Day 1 (tetanus) | 0.62 [0.5 to 0.76] | 0.75 [0.61 to 0.92]
  Day 29 (tetanus) | 12 [9.84 to 14] | 15 [13 to 18]
  Day 1 (PT ) (N=286,287) | 2.68 [1.97 to 3.66] | 2.85 [2.1 to 3.86]
  Day 29 (PT) (N=286,287) | 62 [52 to 74] | 79 [66 to 93]
  Day 1 (FHA) (N=286,287) | 15 [13 to 18] | 17 [14 to 20]
  Day 29 (FHA) (N=286,287) | 186 [165 to 209] | 219 [194 to 246]
  Day 1 (PRN) (N=285,287) | 6.45 [5.18 to 8.03] | 8.7 [7.01 to 11]
  Day 29 (PRN) (N=285,287) | 157 [131 to 189] | 254 [211 to 304]

4. Secondary Outcome: Geometric Mean Ratios of Antibody Concentrations Against Diphtheria,Tetanus and Pertussis Antigens When Tdap is Administered Concomitantly With MenACWY-CRM Vaccine Compared to Tdap Given Concomitantly With Saline Placebo
Description: The geometric mean ratios (GMRs- day 29/day 1) of post-vaccination versus pre- vaccination antibody concentrations against diptheria, tetanus and pertussis (PT, FHA and PRN) antigens following concomitant administration of Tdap vaccine with MenACWY-CRM vaccine as compared to when Tdap was given concomitantly with saline placebo.
Time Frame: 1 month after vaccination (Day 29)
Population: Analysis was done on per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Tdap+ MenACWY-CRM | Tdap+Saline
Number analyzed (Participants) | 350 | 345
Ratio
  diphtheria | 72 [58 to 91] | 22 [18 to 28]
  tetanus | 19 [14 to 25] | 20 [15 to 26]
  PT (N=286,287) | 23 [18 to 30] | 28 [21 to 36]
  FHA (N=286,287) | 12 [10 to 14] | 13 [11 to 15]
  PRN (N=285,287) | 24 [20 to 30] | 29 [24 to 35]

5. Secondary Outcome: Percentage of Subjects With Serum Bactericidal Antibody Titers ≥1:4 and ≥1:8, When MenACWY-CRM is Concomitantly Administered With Tdap Vaccine Compared to MenACWY-CRM Given Concomitantly With Saline Placebo
Description: The percentage of subjects with serum bactericidal antibody titers(hSBA) ≥ 1:4 and ≥ 1:8 against Neisseria meningitidis serogroups A,C,W and Y,following concomitant administration of MenACWY-CRM vaccine with Tdap vaccine as compared to when MenACWY-CRM was given concomitantly with saline placebo.
  The serum bactericidal antibodies directed against N.meningitidis serogroup A, C, W and Y, are measured by human complement Serum Bactericidal Assay (hSBA).
Time Frame: 1 month after vaccination (Day 29)
Population: Analysis was done on per-protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Tdap + MenACWY-CRM | MenACWY-CRM + Saline
Number analyzed (Participants) | 119 | 126
Percentages of subjects
  Day 1 (Men A) hSBA ≥ 1:4 | 3 [1 to 7] | 5 [2 to 10]
  Day 29 (Men A) hSBA ≥ 1:4 | 79 [71 to 86] | 83 [75 to 89]
  Day 1 (Men C) hSBA ≥ 1:4 (N=118,124) | 36 [28 to 46] | 30 [22 to 39]
  Day 29 (Men C) hSBA ≥ 1:4 (N=118,124) | 94 [88 to 98] | 90 [84 to 95]
  Day 1 (Men W) hSBA ≥ 1:4 (N=116,124) | 57 [47 to 66] | 56 [47 to 65]
  Day 29 (Men W) hSBA ≥ 1:4 (N=116,124) | 97 [93 to 99] | 97 [92 to 99]
  Day 1 (Men Y) hSBA ≥ 1:4 (N=117,125) | 47 [38 to 56] | 42 [33 to 51]
  Day 29 (Men Y) hSBA ≥ 1:4 (N=117,125) | 96 [90 to 99] | 97 [92 to 99]
  Day 1 (Men A) hSBA ≥ 1:8 | 2 [0 to 6] | 4 [1 to 9]
  Day 29 (Men A) hSBA ≥ 1:8 | 74 [65 to 82] | 80 [72 to 87]
  Day 1 (Men C) hSBA ≥ 1:8 (N=118,124) | 25 [17 to 33] | 25 [18 to 34]
  Day 29 (Men C) hSBA ≥ 1:8 (N=118,124) | 92 [86 to 96] | 88 [81 to 93]
  Day 1 (Men W) hSBA ≥ 1:8 (N=116,124) | 53 [43 to 62] | 56 [46 to 65]
  Day 29 (Men W) hSBA ≥ 1:8 (N=116,124) | 96 [90 to 99] | 97 [92 to 99]
  Day 1 (Men Y) hSBA ≥ 1:8 (N=117,125) | 38 [30 to 48] | 38 [29 to 47]
  Day 29 (Men Y) hSBA ≥ 1:8 (N=117,125) | 93 [87 to 97] | 94 [89 to 98]

6. Secondary Outcome: The hSBA Geometric Mean Titers Against N.Meningitidis Serogroups A,C,W and Y, When MenACWY-CRM is Concomitantly Administered With Tdap Vaccine Compared to MenACWY-CRM Given Concomitantly With Saline Placebo
Description: The hSBA geometric mean titers (GMTs) against N.meningitidis serogroups A,C,W and Y, at baseline and at one month, following concomitant administration of MenACWY-CRM vaccine with Tdap vaccine, as compared to when MenACWY-CRM was given concomitantly with saline placebo.
Time Frame: 1 month after vaccination (Day 29)
Population: Analysis was done on per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Tdap + MenACWY-CRM | MenACWY-CRM + Saline
Number analyzed (Participants) | 119 | 126
Titers
  Day 1 (Men A) | 2.14 [1.99 to 2.31] | 2.21 [2.05 to 2.38]
  Day 29 (Men A) | 34 [23 to 50] | 50 [34 to 74]
  Day 1 (Men C) N=118,124 | 4 [3.23 to 4.96] | 3.92 [3.16 to 4.86]
  Day 29 (Men C) N=118,124 | 89 [58 to 136] | 92 [60 to 140]
  Day 1 (Men W) N=116,124 | 11 [7.7 to 15] | 9.49 [6.93 to 13]
  Day 29 (Men W) N=116,124 | 73 [54 to 98] | 77 [57 to 103]
  Day 1 (Men Y) N=117,125 | 5.38 [4.2 to 6.89] | 5 [3.91 to 6.39]
  Day 29 (Men Y) N=117,125 | 73 [54 to 98] | 70 [52 to 94]

7. Secondary Outcome: Geometric Mean Ratios of hSBA Titers Against N.Meningitidis Serogroups A,C,W and Y, When MenACWY-CRM is Concomitantly Administered With Tdap Compared to MenACWY-CRM Given Concomitantly With Saline Placebo
Description: The geometric mean ratios (GMRs-day 29/day1)of post-vaccination versus pre- vaccination hSBA titers against N.meningitidis serogroups A,C,W and Y, when MenACWY-CRM vaccine is concomitantly administered with Tdap vaccine as compared to when MenACWY-CRM was given concomitantly with saline placebo.
Time Frame: 1 month after vaccination (Day 29)
Population: Analysis was done on per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | Tdap + MenACWY-CRM | MenACWY-CRM + Saline
Number analyzed (Participants) | 119 | 126
Ratios
  Men A | 16 [11 to 23] | 23 [16 to 33]
  Men C (N=118,124) | 22 [15 to 33] | 23 [16 to 35]
  Men W (N=116,124) | 6.9 [4.84 to 9.85] | 8.09 [5.69 to 12]
  Men Y (N=117,125) | 14 [9.41 to 19] | 14 [9.79 to 20]

8. Secondary Outcome: Percentage of Subjects With hSBA Seroresponse, When MenACWY-CRM is Concomitantly Administered With Tdap Compared to MenACWY-CRM Given Concomitantly With Saline Placebo
Description: The percentage of subjects showing an hSBA seroresponse against N.meningitidis serogroups A,C,W and Y, following concomitant administration of MenACWY-CRM vaccine with Tdap vaccine as compared to when MenACWY-CRM was given concomitantly with saline placebo.
  Seroresponse to MenACWY-CRM is defined as a pre-vaccination hSBA titer < 1:4 to a post-vaccination hSBA titer of ≥ 1:8 or a pre-vaccination hSBA titer ≥ 1:4 to a post-vaccination titer of at least four times the baseline hSBA titer.
Time Frame: 1 month after vaccination (Day 29)
Population: Analysis was done on per-protocol population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Tdap + MenACWY-CRM | MenACWY-CRM + Saline
Number analyzed (Participants) | 119 | 126
Percentages of subjects
  Men A | 74 [65 to 82] | 80 [72 to 87]
  Men C (N=118, 124) | 82 [74 to 89] | 78 [70 to 85]
  Men W (N=116, 124) | 58 [48 to 67] | 59 [50 to 68]
  Men Y (N=117, 125) | 70 [61 to 78] | 70 [61 to 78]

9. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Adverse Events When Tdap is Concomitantly Administered With MenACWY-CRM Compared to When MenACWY-CRM is Concomitantly Administered With Saline Placebo
Description: The number of subjects reporting solicited local and systemic reactions following concomitant administration of MenACWY-CRM vaccine and Tdap vaccine as compared to when MenACWY-CRM vaccine was concomitantly administered with saline placebo.
Time Frame: Day 1-7 after any vaccination
Population: Analysis was done on the safety population
Measure: Number; unit: Participants
Arm/Group | Tdap + MenACWY-CRM | MenACWY-CRM + Saline
Number analyzed (Participants) | 359 | 357
Participants
  Local | 278 | 179
  Injection site pain (MenACWY) site 1 | 82 | 116
  Injection site erythema (MenACWY) site 1 | 48 | 66
  Injection site induration (MenACWY) site 1 | 41 | 59
  Injection site pain (Tdap or saline) site 2 | 246 | 57
  Injection site erythema (Tdap or saline) site 2 | 103 | 37
  Injection site induration (Tdap or saline) site 2 | 118 | 23
  Systemic | 198 | 171
  Chills | 39 | 47
  Nausea | 43 | 28
  Malaise | 65 | 43
  Myalgia | 118 | 79
  Arthralgia | 57 | 40
  Headache | 129 | 128
  Fever ≥ 38°C | 11 | 14
  Other | 42 | 33
  Stayed home due to reaction (N=358,357) | 12 | 12
  Analgesic Antipyretic medication used | 38 | 31

10. Secondary Outcome: Number of Subjects With Solicited Local and Systemic Adverse Events When Tdap is Concomitantly Administered With MenACWY-CRM Compared to When Tdap is Concomitantly Administered With Saline Placebo
Description: The number of subjects reporting solicited local and systemic reactions following concomitant administration of MenACWY-CRM vaccine and Tdap vaccine as compared to when Tdap was concomitantly administered with saline placebo
Time Frame: Day 1-7 after any vaccination
Population: Analysis was done on the safety population
Measure: Number; unit: Participants
Arm/Group | Tdap + MenACWY-CRM | Tdap + Saline
Number analyzed (Participants) | 359 | 353
Participants
  Local | 278 | 282
  Injection site pain (Tdap) site 2 | 227 | 246
  Injection site erythema (Tdap) site 2 | 103 | 103
  Injection site induration (Tdap) site 2 | 110 | 118
  Injection site pain (MenACWY or saline) site 1 | 82 | 41
  Injection site erythema (MenACWY or saline) site 1 | 48 | 34
  Injection site induration(MenACWY or saline)site1 | 41 | 27
  Systemic | 198 | 202
  Chills | 39 | 41
  Nausea | 43 | 35
  Malaise | 65 | 57
  Myalgia | 118 | 127
  Arthralgia | 57 | 60
  Headache | 129 | 110
  Fever ≥ 38°C | 11 | 7
  Other | 42 | 39
  Stayed home due to reaction (N=358,353) | 12 | 15
  Analgesic Antipyretic medication used | 38 | 38

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events When Tdap is Concomitantly Administered With MenACWY-CRM Compared to MenACWY-CRM or Tdap Concomitantly Administered With Saline Placebo
Description: The number of subjects reporting any unsolicited adverse events (AEs) when Tdap is concomitantly administered with MenACWY-CRM as compared to when MenACWY-CRM vaccine or Tdap vaccine was concomitantly administered with saline placebo.
Time Frame: Throughout the study (Day 1 to Day 181)
Population: This analysis was done on the safety population.
Measure: Number; unit: Participants
Arm/Group | Tdap + MenACWY-CRM | Tdap + Saline | MenACWY-CRM + Saline
Number analyzed (Participants) | 359 | 353 | 357
Participants
  Any AE (Day 1 to 29) | 43 | 31 | 48
  Possibly/probably related AE (Day 1 to 29) | 8 | 6 | 6
  Serious AEs (Day 1 to 29) | 0 | 0 | 0
  AE's leading to discontinuation (Day 1 to 29) | 0 | 0 | 0
  Possibly/probably related SAE(Day 1 to 29) | 0 | 0 | 0
  Death ( Day 1 to 29) | 0 | 0 | 0
  Any AE (Day 30 to 181) | 42 | 36 | 39
  Possibly/probably related AE (Day 30 to 181) | 0 | 0 | 0
  Serious AEs (Day 30 to 181) | 1 | 2 | 0
  AE's leading to discontinuation (Day 30 to 181) | 0 | 0 | 0
  Possibly/probably related SAE (Day 30 to 181) | 0 | 0 | 0
  Death (Day 30 to 181) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All serious adverse events were collected throughout the study (Day 1-181). All solicited events were collected from Day 1-7 post vaccination; unsolicited adverse events were collected from Day 1-181.
Description: There were 3 subjects who withdrew consent (2 subjects in the Tdap+MenACWY-CRM group and 1 subject in the Tdap+Saline group) prior to visit one of the study and thus were not included in the safety analyses for this section.
Arm/Group | Tdap + MenACWY-CRM | Tdap + Saline | MenACWY-CRM + Saline
Serious Adverse Events (participants affected / at risk) | 1/359 | 2/353 | 0/357
Other Adverse Events (participants affected / at risk) | 297/359 | 309/353 | 238/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tdap + MenACWY-CRM (N=359) | Tdap + Saline (N=353) | MenACWY-CRM + Saline (N=357)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tdap + MenACWY-CRM (N=359) | Tdap + Saline (N=353) | MenACWY-CRM + Saline (N=357)
Nausea (Gastrointestinal disorders) | 44 | 38 | 31
Chills (General disorders) | 39 | 41 | 47
Injection site erythema (General disorders) | 119 | 110 | 83
Injection site induration (General disorders) | 125 | 131 | 72
Injection site pain (General disorders) | 259 | 262 | 139
Malaise (General disorders) | 67 | 57 | 43
Pyrexia (General disorders) | 21 | 14 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 60 | 40
Myalgia (Musculoskeletal and connective tissue disorders) | 119 | 128 | 80
Headache (Nervous system disorders) | 131 | 113 | 136

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days